CLINICAL TRIAL: NCT00441337
Title: A Phase 1, Open Label, Dose-escalation, Safety and Pharmacokinetic Study of MDX-1106 in Patients With Selected or Relapsed Malignancies
Brief Title: A Study of MDX-1106 in Patients With Selected Refractory or Relapsed Malignancies
Acronym: MDX1106-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-001 ST; MDX1106-01 (Other: BMS)
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Results first posted 2015-02-20 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Colorectal Cancer; Malignant Melanoma; Renal Cancer; Prostate Cancer
Keywords: malignancies; cancer; non small cell lung cancer; lung cancer; colorectal cancer; adenocarcinoma; melanoma; malignant melanoma; renal cancer; renal carcinoma; carcinoma; prostate cancer; prostate adenocarcinoma; Recurrent or treatment refractory malignancies
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Melanoma; Kidney Neoplasms; Prostatic Neoplasms; Neoplasms; Lung Neoplasms; Adenocarcinoma; Carcinoma, Renal Cell; Carcinoma; Recurrence | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.3 mg/kg MDX-1106 drug (Experimental): 0.3 milligrams (mg) MDX-1106 drug (nivolumab) per kilogram (kg) of body weight (mg/kg) was administered in a single intravenous (IV) infusion. If criteria were met, 2 additional doses could be administered (1 every 4 weeks).
  Interventions: Biological: MDX-1106
- 1 mg/kg MDX-1106 drug (Experimental): 1 mg MDX-1106 drug (nivolumab) per kg of body weight (mg/kg) was administered in a single IV infusion. If criteria were met, 2 additional doses could be administered (1 every 4 weeks).
  Interventions: Biological: MDX-1106
- 3 mg/kg MDX-1106 drug (Experimental): 3 mgs MDX-1106 drug (nivolumab) per kg of body weight (mg/kg) was administered in a single IV infusion. If criteria were met, 2 additional doses could be administered (1 every 4 weeks).
  Interventions: Biological: MDX-1106
- 10 mg/kg MDX-1106 drug (Experimental): 10 mgs MDX-1106 drug (nivolumab) per kg of body weight (mg/kg) was administered in a single IV infusion. If criteria were met, 2 additional doses could be administered (1 every 4 weeks).
  Interventions: Biological: MDX-1106

INTERVENTIONS:
Biological: MDX-1106 — patients will receive a single dose of MDX-1106 as a 60 minute infusion.
  Other Names: nivolumab

SUMMARY:
To evaluate the safety, tolerability, efficacy, and pharmacokinetics of MDX-1106 when administered to patients with advanced non-small cell lung cancer, colorectal cancer, malignant melanoma, clear cell renal cell cancer or hormone refractory prostate cancer

DETAILED DESCRIPTION:
Six patients enrolled at each dose level of 0.3, 1.0, 3.0 and 10mg/kg; the remaining 10 to 15 patients may subsequently be enrolled at a dose at or below the maximum tolerated dose (MTD) during the dose-escalation portion of the study. Patients who respond may receive additional doses of drug.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed/refractory non-small cell lung cancer, colorectal adenocarcinoma, malignant melanoma, renal (clear) cell carcinoma, or hormone-refractory prostate adenocarcinoma
* Prior treatment must have been completed at least 4 weeks prior to enrollment
* No untreated primary or metastatic brain or meningeal tumors
* ECOG PS 0 or 1
* Meet all screening laboratory values

Exclusion Criteria:

* History of severe hypersensitivity reactions to other monoclonal antibodies
* Active autoimmune disease or a documented history of autoimmune disease
* Prior therapy with an anti-PD-1 or anti-CTLA-4 antibody
* Active infection
* Concurrent medical condition requiring the use of immunosuppressive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - Johns Hopkins Unv., School of Medicine, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine - Barnes Jewish Hospital, St Louis, Missouri
  - Carolina BioOncology Institute, PLLC, Huntersville, North Carolina

REFERENCES:
- [Derived] George S, Pili R, Carducci MA, Kim JJ. Role of immunotherapy for renal cell cancer in 2011. J Natl Compr Canc Netw. 2011 Sep 1;9(9):1011-8. doi: 10.6004/jnccn.2011.0085. PMID 21917625

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study from 25 October 2006 to 27 November 2009. After completion of a single dose (cycle 1), those meeting criteria could be re-treated with 2 additional doses (cycle 2); and additional cycles. Participants who had a complete response (CR) or partial response (PR) at end of re-treatment were followed-up until disease progression for 2 years.
Pre-assignment Details: 39 participants were enrolled and 39 were treated with at least 1 dose or a partial dose of study drug.
Groups:
- 0.3 mg/kg Nivolumab: 0.3 milligrams (mg) of nivolumab per kilogram (kg) of body weight (mg/kg) was administered in a single intravenous (IV) infusion on Day 1 with 10% of the dose infused over 6 minutes and after a 1 hour observation period, the balance was administered over 60 minutes. Eligible participants could be re-treated and receive 2 more doses (1 dose every 4 weeks) at same dose as the single dose if: disease was stable, no drug intolerance was observed, no complete response (CR) or partial response (PR) was observed, or they had a positive immunogenicity sample within 4 weeks prior to re-treatment. Those who responded to therapy with a CR or PR were eligible for long-term follow-up until either progressive disease (PD) or 2 years elapsed.
- 1 mg/kg Nivolumab: 1 mg of nivolumab per kg of body weight was administered in a single IV infusion over 60 minutes on Day 1. Eligible participants could be re-treated and receive 2 more doses (1 dose every 4 weeks) at same dose as the single dose if: disease was stable, no drug intolerance was observed, no complete response (CR) or partial response (PR) was observed, or they had a positive immunogenicity sample within 4 weeks prior to re-treatment. Those who responded to therapy with a CR or PR were eligible for long-term follow-up until either progressive disease (PD) or 2 years elapsed.
- 3 mg/kg Nivolumab: 3 mg of nivolumab per kg of body weight was administered in a single IV infusion over 60 minutes on Day 1. Eligible participants could be re-treated and receive 2 more doses (1 dose every 4 weeks) at same dose as the single dose if: disease was stable, no drug intolerance was observed, no complete response (CR) or partial response (PR) was observed, or they had a positive immunogenicity sample within 4 weeks prior to re-treatment. Those who responded to therapy with a CR or PR were eligible for long-term follow-up until either progressive disease (PD) or 2 years elapsed.
- 10 mg/kg Nivolumab: 10 mg of nivolumab per kg of body weight was administered in a single IV infusion over 60 minutes on Day 1. Eligible participants could be re-treated and receive 2 more doses (1 dose every 4 weeks) at same dose as the single dose if: disease was stable, no drug intolerance was observed, no complete response (CR) or partial response (PR) was observed, or they had a positive immunogenicity sample within 4 weeks prior to re-treatment. Those who responded to therapy with a CR or PR were eligible for long-term follow-up until either progressive disease (PD) or 2 years elapsed.
Period: Overall Study
Arm/Group | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Started | 6 | 6 | 6 | 21
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 6 | 21
Not completed — Disease Progression | 6 | 6 | 4 | 18
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Sponsor Decision | 0 | 0 | 1 | 2
Not completed — Did not meet inclusion criteria | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose or any partial dose of study drug.
Groups:
- 0.3 mg/kg Nivolumab: 0.3 mg of nivolumab per kg of body weight (mg/kg) was administered in a single IV infusion on Day 1 with 10% of the dose infused over 6 minutes and after a 1 hour observation period, the balance was administered over 60 minutes. Eligible participants could be re-treated and receive 2 more doses (1 dose every 4 weeks) at same dose as the single dose if: disease was stable, no drug intolerance was observed, no complete response (CR) or partial response (PR) was observed, or they had a positive immunogenicity sample within 4 weeks prior to re-treatment. Those who responded to therapy with a CR or PR were eligible for long-term follow-up until either progressive disease (PD) or 2 years elapsed.
- Total: Total of all reporting groups
Arm/Group | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab | Total
Number analyzed (Participants) | 6 | 6 | 6 | 21 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (5.7) | 68.3 (9.4) | 61.0 (10.4) | 63.2 (10.0) | 62.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 10 | 17
  Male | 4 | 3 | 4 | 11 | 22
Race/Ethnicity, Customized [Number; unit: participants]
  White | 4 | 3 | 4 | 18 | 29
  Black | 2 | 3 | 2 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 21 | 39
Body Weight in kilograms (kg) [Median (Full Range); unit: kg] | 96.8 [88 to 136] | 73.9 [62 to 80] | 81.9 [55 to 98] | 81.3 [56 to 118] | 81.3 [55 to 136]
Time since initial diagnosis (years) [Median (Full Range); unit: Years] | 3.7 [1.4 to 6.8] | 2.7 [1.5 to 14.0] | 5.6 [0.7 to 11.4] | 4.1 [1.0 to 19.8] | 3.8 [0.7 to 19.8]
Type of Malignancy [Number; unit: participants]
  Prostate Cancer | 0 | 1 | 2 | 5 | 8
  Melanoma | 0 | 2 | 0 | 8 | 10
  Non-small cell lung cancer | 1 | 1 | 2 | 2 | 6
  Renal cell cancer | 0 | 0 | 0 | 1 | 1
  Colorectal cancer | 5 | 2 | 2 | 5 | 14
Stage of Malignancy at Screening Diagnosis [Number; unit: participants] — The investigator reported the screening malignancy stage for each type of cancer using the American Joint Committee on Cancer Classification (Stages I, II, III, and IV).
  participants
    Stage I | 0 | 0 | 0 | 0 | 0
    Stage II | 0 | 0 | 0 | 0 | 0
    Stage III | 1 | 0 | 0 | 0 | 1
    Stage IV | 5 | 6 | 6 | 21 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Severe Adverse Events (AEs), Serious Adverse Events (SAEs), Drug-Related AEs, Deaths, Discontinuation of Study Drug Due to AE, Dose-Limiting Toxicity (DLT) AE and Immune-related AEs (irAEs) in Safety Population
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling. Severe=All Grade 3 or 4 events. Death=during the study and up to 28 days past study discontinuation. AEs graded using the Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0. irAEs=unknown etiology, associated with study drug and consistent with an immune phenomenon. DLT: ≥Gr 3 AE(s) or lab abnormality without alternative explanation other than drug.
Time Frame: Day 1 to 70 days post last dose of study drug; 28 days past study discontinuation
Population: Safety Population: All participants who received at least 1 dose or any partial dose of nivolumab were analyzed.
Measure: Number; unit: participants
Arm/Group | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 6 | 6 | 6 | 21
participants
  Severe AE | 5 | 5 | 4 | 18
  SAE | 3 | 5 | 4 | 9
  SAE through 28 days post study discontinuation | 3 | 5 | 4 | 11
  Drug-Related AE | 5 | 5 | 6 | 19
  Death | 1 | 4 | 1 | 6
  Discontinuation of Study Drug due to AE | 0 | 0 | 0 | 2
  irAE | 1 | 3 | 2 | 9
  Dose-Limiting Toxicity AE | 0 | 0 | 0 | 0

2. Primary Outcome: Geometric Mean Maximum Serum Concentration (Cmax) Observed Post-Single Dose
Description: Nivolumab in human serum was assayed during the period of known analyte stability and reported as final data for this study by PPD® (Richmond, Virginia) using a cross-validated enzyme-linked immunosorbent assay (ELISA) method. For the single dose (Day 1), serum concentrations of nivolumab were assessed: prior to dosing, at 30 minutes (during dosing), immediately post-dose, and 30 minutes post-infusion end time; at 1, 2, 4, 6, 8, 24, 48, and 72 hours post-infusion end time; and on Days 8, 15, 22, 29, 43, 57, 71, and 85. The pharmacokinetic (PK) parameter of Cmax was measured in micrograms per milliliter (µg/mL).
Time Frame: Day 1 to Day 85
Population: All participants who received at least 1 dose or any partial dose of nivolumab and had adequate PK profiles were included in the summary statistics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- 0.3 mg/kg Nivolumab: 0.3 mg of nivolumab per kg of body weight (mg/kg) was administered in a single IV infusion on Day 1 with 10% of the dose infused over 6 minutes and after a 1 hour observation period, the balance was administered over 60 minutes. Eligible participants could be re-treated and receive 2 more doses (1 dose every 4 weeks) at same dose as the single dose if: disease was stable, no drug intolerance was observed, no CR or PR was observed, or they had a positive immunogenicity sample within 4 weeks prior to re-treatment. Those who responded to therapy with a CR or PR were eligible for long-term follow-up until either PD or 2 years elapsed.
- 1 mg/kg Nivolumab: 1 mg of nivolumab per kg of body weight was administered in a single IV infusion over 60 minutes on Day 1. Eligible participants could be re-treated and receive 2 more doses (1 dose every 4 weeks) at same dose as the single dose if: disease was stable, no drug intolerance was observed, no CR or PR was observed, or they had a positive immunogenicity sample within 4 weeks prior to re-treatment. Those who responded to therapy with a CR or PR were eligible for long-term follow-up until either PD or 2 years elapsed.
- 3 mg/kg Nivolumab: 3 mg of nivolumab per kg of body weight was administered in a single IV infusion over 60 minutes on Day 1. Eligible participants could be re-treated and receive 2 more doses (1 dose every 4 weeks) at same dose as the single dose if: disease was stable, no drug intolerance was observed, no CR or PR was observed, or they had a positive immunogenicity sample within 4 weeks prior to re-treatment. Those who responded to therapy with a CR or PR were eligible for long-term follow-up until either PD or 2 years elapsed.
- 10 mg/kg Nivolumab: 10 mg of nivolumab per kg of body weight was administered in a single IV infusion over 60 minutes on Day 1. Eligible participants could be re-treated and receive 2 more doses (1 dose every 4 weeks) at same dose as the single dose if: disease was stable, no drug intolerance was observed, no CR or PR was observed, or they had a positive immunogenicity sample within 4 weeks prior to re-treatment. Those who responded to therapy with a CR or PR were eligible for long-term follow-up until either PD or 2 years elapsed.
Arm/Group | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 6 | 6 | 5 | 21
µg/mL | 6.7 (21.6) | 16.0 (32.1) | 60.0 (27.6) | 196.3 (19.5)

3. Primary Outcome: Median Time at Which the Maximum Serum Concentration Occurred (Tmax) Post-Single Dose
Description: Nivolumab in human serum was assayed during the period of known analyte stability and reported as final data for this study by PPD® (Richmond, Virginia) using a cross-validated ELISA method. For the single dose (Day 1), serum concentrations of nivolumab were assessed: prior to dosing, at 30 minutes (during dosing), immediately post-dose, and 30 minutes post-infusion end time; at 1, 2, 4, 6, 8, 24, 48, and 72 hours post-infusion end time; and on Days 8, 15, 22, 29, 43, 57, 71, and 85. The PK parameter of Tmax was measured in hours (h).
Time Frame: Day 1 to Day 85
Population: as for outcome 2
Measure: Median (Full Range); unit: h
Arm/Group | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 6 | 6 | 5 | 21
h | 3.0 [1.0 to 6.8] | 1.9 [1.0 to 7.0] | 3.1 [1.0 to 5.0] | 1.6 [0.9 to 7.0]

4. Primary Outcome: Geometric Mean Area Under the Curve (AUC) From Time of Dosing to Time of Last Observation (0-T) and Extrapolated to Infinity (INF) Observed Post-Single Dose
Description: AUC(0-T): Area under the concentration-time curve from the time of dosing to the time of the last observation. AUC(INF): Area under the curve from the time of dosing extrapolated to infinity. Nivolumab in human serum was assayed during the period of known analyte stability and reported as final data for this study by PPD® (Richmond, Virginia) using a cross-validated ELISA method. For the single dose (Day 1), serum concentrations of nivolumab were assessed: prior to dosing, at 30 minutes (during dosing), immediately post-dose, and 30 minutes post-infusion end time; at 1, 2, 4, 6, 8, 24, 48, and 72 hours post-infusion end time; and on Days 8, 15, 22, 29, 43, 57, 71, and 85. The PK parameters of AUC(0-T) and AUC (INF) were measured in micrograms*hours per milliliter (µg*h/mL).
Time Frame: Day 1 to Day 85
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Groups:
- 0.3 mg/kg Nivolumab: 0.3 mg of nivolumab per kg of body weight was administered in a single IV infusion on Day 1 with 10% of the dose infused over 6 minutes and after a 1 hour observation period, the balance was administered over 60 minutes. Eligible participants could be re-treated and receive 2 more doses (1 dose every 4 weeks) at same dose as the single dose if: disease was stable, no drug intolerance was observed, no CR or PR was observed, or they had a positive immunogenicity sample within 4 weeks prior to re-treatment. Those who responded to therapy with a CR or PR were eligible for long-term follow-up until either PD or 2 years elapsed.
Arm/Group | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 6 | 6 | 5 | 21
µg*h/mL
  AUC (0-T); n=6, 6, 5, 21 | 970 (47) | 3244 (62) | 13909 (44) | 55324 (39)
  AUC (INF); n=3, 4, 5, 19 | 2343 (16) | 6014 (30) | 15813 (44) | 76541 (27)

5. Primary Outcome: Mean Elimination Half-life (T-HALF) Post-Single Dose
Description: Nivolumab in human serum was assayed during the period of known analyte stability and reported as final data for this study by PPD® (Richmond, Virginia) using a cross-validated ELISA method. For the single dose (Day 1), serum concentrations of nivolumab were assessed: prior to dosing, at 30 minutes (during dosing), immediately post-dose, and 30 minutes post-infusion end time; at 1, 2, 4, 6, 8, 24, 48, and 72 hours post-infusion end time; and on Days 8, 15, 22, 29, 43, 57, 71, and 85. The PK parameter of T-HALF was measured in days.
Time Frame: Day 1 to Day 85
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 3 | 4 | 5 | 19
days | 18.9 (7.05) | 17.0 (2.36) | 17.0 (4.70) | 24.8 (7.22)

6. Primary Outcome: Geometric Mean Total Body Clearance of Drug From Serum (CLT) Post-Single Dose
Description: Nivolumab in human serum was assayed during the period of known analyte stability and reported as final data for this study by PPD® (Richmond, Virginia) using a cross-validated ELISA method. For the single dose (Day 1), serum concentrations of nivolumab were assessed: prior to dosing, at 30 minutes (during dosing), immediately post-dose, and 30 minutes post-infusion end time; at 1, 2, 4, 6, 8, 24, 48, and 72 hours post-infusion end time; and on Days 8, 15, 22, 29, 43, 57, 71, and 85. The PK parameter of CLT was measured in milliliters per hour per kilogram body weight (mL/h/kg).
Time Frame: Day 1 to Day 85
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h/kg
Arm/Group | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 3 | 4 | 5 | 19
mL/h/kg | 0.13 (16.93) | 0.17 (29.80) | 0.19 (42.66) | 0.13 (28.42)

7. Primary Outcome: Mean Volume of Distribution (Vz) Post-Single Dose
Description: Nivolumab in human serum was assayed during the period of known analyte stability and reported as final data for this study by PPD® (Richmond, Virginia) using a cross-validated ELISA method. For the single dose (Day 1), serum concentrations of nivolumab were assessed: prior to dosing, at 30 minutes (during dosing), immediately post-dose, and 30 minutes post-infusion end time; at 1, 2, 4, 6, 8, 24, 48, and 72 hours post-infusion end time; and on Days 8, 15, 22, 29, 43, 57, 71, and 85. The PK parameter of Vz was measured in milliliters per kilogram of body weight (mL/kg).
Time Frame: Day 1 to Day 85
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 3 | 4 | 5 | 19
mL/kg | 82.8 (27.19) | 99.6 (23.04) | 112.7 (39.50) | 109.4 (26.70)

8. Primary Outcome: Percent of Participants With Best Overall Response Rate in Safety Population and in Tumor Evaluable Population
Description: The Best Overall Response Rate (BORR) was defined as the number of participants who had a confirmed complete response (CR) or partial response (PR) during the study divided by the total number of participants evaluated. Response was based on tumor assessment for both target and non-target lesions using: Clinical examination; Chest X-ray; Computed Tomography and Magnetic Resonance Imaging; Bone scan; Ultrasound. Per National Cancer Institute Response Evaluation Criteria in Solid Tumors (RECIST) v1.0, best overall response (BOR) for tumors was confirmed CR or PR. CR=disappearance of all target and non-target lesions; PR=at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the screening sum longest diameter. Confidence intervals (CIs) were computed using the Clopper and Pearson method.
Time Frame: Day 1 up to 2 Years.
Population: Safety Population: All participants who received at least 1 dose or any partial dose of nivolumab were analyzed. Tumor Evaluable Population: all participants who received complete dose(s) of nivolumab and had completed a major tumor assessment (a baseline and at least 1 post-baseline tumor assessment for either target and/or non-target assessments.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 6 | 6 | 6 | 21
percentage of participants
  Safety Population (n=6,6,6,21) | 0 [0.0 to 45.9] | 0 [0.0 to 45.9] | 16.7 [0.4 to 64.1] | 9.5 [1.2 to 30.4]
  Tumor Evaluable Population (n=6,5,6,20) | 0 [0.0 to 45.9] | 0 [0.0 to 52.2] | 16.7 [0.4 to 64.1] | 10.0 [1.2 to 31.7]

9. Primary Outcome: Percent of Participants With Prostate-Specific Antigen (PSA) Response After the First Dose by Day 85 In Participants With Hormone-Refractory Prostate Adenocarcinoma (HRPC)
Description: The PSA response rate was defined as the number of participants who had at least a 50% decrease of the PSA value from the PSA reference value divided by the total number of participants evaluated (percent of participants). PSA reference value was the PSA concentration measured immediately prior to dosing on Day 1. PSA response was assessed using the Recommendations from the National Cancer Institute Prostate-Specific Antigen Working Group. A PSA response had to be confirmed at least 4 weeks after first response. 95% exact CIs were computed using the Clopper and Pearson method.
Time Frame: Day 1 to Day 85
Population: The PSA evaluable population was analyzed and included all HRPC participants who received complete dose(s) of nivolumab and had a baseline PSA assessment and at least one post baseline PSA assessment. A PSA evaluable participant could not have any major inclusion/exclusion violation, dosing violation, or protocol conduct violation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 0 | 1 | 2 | 5
percentage of participants |  | 0 [0.0 to 97.5] | 0 [0.0 to 84.2] | 0 [0.0 to 52.2]

10. Secondary Outcome: Number of Participants With Best Overall Response (BOR) by Category in Safety Population
Description: Measurable and non-measurable disease/target lesions were evaluated according to National Cancer Institute standardized RECIST.Complete Response (CR)=disappearance of all target and non-target lesions and no new lesions; Partial Response=at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the screening sum longest diameter; Stable disease (SD)=neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum longest diameter since treatment; PD=at least a 20% increase in the sum of the longest diameter recorded since screening, or the appearance of one or more new lesions. BOR was recorded between the first tumor assessment and last tumor assessment. CR and PR had to be confirmed by repeat assessment no less than 4 weeks after the criteria were first met. SD assessment must have met the criteria at least once at or after Week 12.
Time Frame: Day 1 to Day 85
Population: Safety Population: All participants who received at least 1 dose or any partial dose of nivolumab were analyzed.
Measure: Number; unit: participants
Arm/Group | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 6 | 6 | 6 | 21
participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 1 | 2
  Stable Disease | 1 | 1 | 2 | 6
  Progressive Disease | 5 | 4 | 3 | 12
  Unknown | 0 | 0 | 0 | 1
  Missing | 0 | 1 | 0 | 0

11. Secondary Outcome: Percentage of Participants With Disease Control and Major Durable Disease Control
Description: Disease control rate was defined as number of participants whose Best Overall Response (BOR) was complete response (CR), partial response (PR), or stable disease (SD) divided by the total number of participants. Major durable disease control rate was defined as the total number of participants whose BOR was CR, PR, or SD ≥24 weeks, divided by the total number of participants. Per RECIST v 1.0, BOR for tumors was confirmed CR or PR. CR=disappearance of all target and non-target lesions; PR=at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the screening sum longest diameter since treatment; SD=neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for PD. PD=at least a 20% increase in the sum of the longest diameter recorded since screening, or the appearance of one or more new lesions. 95% CIs were computed using the Clopper and Pearson method.
Time Frame: Day 1 to 2 Years
Population: Safety Population was analyzed: All participants who received at least 1 dose or any partial dose of nivolumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 6 | 6 | 6 | 21
percentage of participants
  Disease Control Rate | 16.7 [0.4 to 64.1] | 16.7 [0.4 to 64.1] | 50.0 [11.8 to 88.2] | 38.1 [18.1 to 61.6]
  Major Durable Disease Control Rate ≥24 weeks | 0 [0.0 to 45.9] | 16.7 [0.4 to 64.1] | 33.3 [4.3 to 77.7] | 4.8 [0.1 to 23.8]

12. Secondary Outcome: Median Time to Tumor Response and Duration of Tumor Response
Description: Time to tumor response: from the date of first dose to the first date of tumor response (CR or PR confirmed at least 4 weeks later); for nonresponders, it was censored at the date of the maximum tumor assessment time in the dose cohort by the end of study. Duration of tumor response was calculated from the first date of response of CR or PR to the date of the first PD or the date of death if a participant died due to disease progression (whichever occurred first). Duration of response was censored at the last tumor assessment date by the end of study if a responder did not have PD or death. Nonresponders had the duration of response as an event of 0 days.
Time Frame: Day 1 to 2 Years
Population: All participants who received at least 1 dose or any partial dose of nivolumab and were tumor responders were analyze.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 0 | 0 | 1 | 2
days
  Time to Tumor Response |  |  | 57 [NA to NA] — insufficient number of participants to calculate CI | 386 [85 to 687]
  Duration of Tumor Response |  |  | 796 [NA to NA] — insufficient number of participants to calculate CI | 327 [92 to 562]

13. Secondary Outcome: Time to Tumor Progression and Tumor Progression Free Survival
Description: Time to tumor progression (TTP) was measured in days from date of the first dose to the date of the first PD or the date of death if due to PD. For those who died without PD it was censored at the date of death. TTP was censored at the last tumor assessment by the end of study if a participant did not have PD or death. Tumor progression free survival (PFS) was measured in days from the date of first dose to the date of the first disease progression or to the date of death. PFS was censored at the last tumor assessment date by the end of study if a participant did not have PD or death.
Time Frame: Day 1 to 2 Years
Population: All participants who received at least 1 dose or any partial dose of nivolumab were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 6 | 6 | 6 | 21
days
  Time to Tumor Progression | 56 [51 to 57] | 57.5 [57 to 59] | 86 [57 to 193] | 57 [53 to 85]
  Tumor Progression Free Survival | 56 [51 to 57] | 57.5 [57 to 59] | 86 [57 to 193] | 57 [53 to 85]

14. Secondary Outcome: Median Time to PSA Progression in Days and Median PSA Progression Free Survival in Days in PSA Evaluable Population
Description: Time to PSA progression: first dose to first PSA progression. Missing date of progression was censored: if death during the study, time to progression was right-censored at last PSA assessment; if no progression from first dose and still alive at end of study, time to progression was right-censored at last PSA assessment by end of study; if no PSA progression and one has discontinued from the study (other than death or PSA progression), time to progression was right-censored at last PSA assessment. PSA progression free survival (PFS): first dose to first PSA progression or death, whichever comes first. Missing date of progression was censored: if one did not have PSA progression from first dose and was still alive at end of study, PSA PFS was right-censored at last PSA assessment; if one does not have any progression and discontinued from the study for reasons other than death or progression, PFS was right-censored at last assessment. CI computed using Brookmeyer and Crowley method.
Time Frame: Day 1 to 2 Years
Population: The PSA evaluable population include all participants in the study who received complete dose(s) of nivolumab and had a baseline PSA assessment and at least 1 post-baseline PSA assessment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 0 | 1 | 2 | 5
days
  Time to PSA Progression |  | 29 [NA to NA] — insufficient number of participants to calculate CI | 58.5 [29 to 88] | 29 [22 to 57]
  PSA Progression Free Survival |  | 29 [NA to NA] — insufficient number of participants to calculate CI | 58.5 [29 to 88] | 29 [22 to 57]

15. Secondary Outcome: Mean Change From Baseline in PSA Relative Velocity at Days 29, 57, and 85 With Cycle 1 in PSA Evaluable Population
Description: PSA relative velocity (PSA RV) was defined as = (d[PSA]/dt)/ [PSA], where [PSA] =concentration of PSA, and t= time, and in the limit reflects the instantaneous change in PSA levels as a fraction of total PSA level. Decreases in PSA RV may occur while measured [PSA] is still rising, and may indicate that continued therapy may lead to a treatment benefit, particularly in the setting of immunotherapy, where expansion of an effective immune response is likely to require weeks to mature. Baseline PSA RV was based on the velocity of last PSA measurement before the first infusion of study drug and the screening PSA measurement.
Time Frame: Day 29, Day 57, Day 85
Population: The PSA evaluable population includes all participants in the study who received complete dose(s) of nivolumab and has a baseline PSA assessment and at least 1 post-baseline PSA assessment.
Measure: Median (Full Range); unit: percentage of total PSA level
Arm/Group | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 0 | 1 | 2 | 5
percentage of total PSA level
  Cycle 1 Day 29 (n=0, 1, 2, 5) |  | 0.009 [0.009 to 0.009] | -0.007 [-0.017 to 0.003] | -0.015 [-0.040 to 0.002]
  Cycle 1 Day 57 (n=0, 1, 2, 5) |  | 0.003 [0.003 to 0.003] | -0.009 [-0.010 to -0.008] | 0.001 [-0.036 to 0.018]
  Cycle 1 Day 85 (n=0, 1, 2, 4) |  | 0.007 [0.007 to 0.007] | 0.001 [-0.003 to 0.004] | -0.005 [-0.044 to 0.017]

16. Secondary Outcome: Mean Change From Baseline in Electrocardiogram Parameters PR, QRS and QT in Safety Population
Description: 12-lead ECGs were performed at screening, baseline, Day 2 and at completion of the dose cycle (Day 85 in first dose cycle). In those participants undergoing re-treatment, ECG was repeated at the completion of the re-treatment. Baseline was defined as the last measurement before the first dose of study drug, which was calculated from pre-dose or from screening if pre-dose was not available. PR, QRS and QT interval were measured in milliseconds (msec).
Time Frame: Baseline, Day 2, Day 85, Day 113
Population: All participants who received at least 1 dose or any partial dose of nivolumab and had available ECG at baseline and on the specified post treatment study day were analyzed.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 6 | 6 | 6 | 21
msec
  PR at Day 2 (n=6,6,6,21) | 7.3 (6.15) | -9.7 (10.31) | -1.7 (9.75) | -0.3 (13.72)
  QRS at Day 2 (n=6,6,6,21) | 5.0 (6.90) | -2.0 (7.48) | -8.7 (19.83) | -1.2 (5.57)
  QT at Day 2 (n=6,6,6,21) | 2.0 (27.86) | -15.7 (22.89) | -2.0 (15.90) | -10.1 (20.76)
  PR at Day 57 (n=0,0,0,3) | NA (NA) — no participants with data on this day in this arm | NA (NA) — no participants with data on this day in this arm | NA (NA) — no participants with data on this day in this arm | -11.3 (24.11)
  QRS at Day 57 (n=0,0,0,3) | NA (NA) — no participants with data on this day in this arm | NA (NA) — no participants with data on this day in this arm | NA (NA) — no participants with data on this day in this arm | 1.3 (5.03)
  QT at Day 57 (n=0,0,0,3) | NA (NA) — no participants with data on this day in this arm | NA (NA) — no participants with data on this day in this arm | NA (NA) — no participants with data on this day in this arm | 5.3 (33.61)
  PR at Day 85 (n=0,4,4,11) | NA (NA) — no participants with data on this day in this arm | -4.5 (11.82) | 3.5 (17.69) | -1.1 (17.44)
  QRS at Day 85 (n=0,4,4,11) | NA (NA) — no participants with data on this day in this arm | -6.0 (9.09) | -4.0 (6.73) | 0.2 (4.24)
  QT at Day 85 (n=0,4,4,11) | NA (NA) — no participants with data on this day in this arm | -6.0 (27.90) | -3.5 (33.52) | -0.2 (26.40)
  PR at Day 113 (n=0,0,2,3) | NA (NA) — no participants with data on this day in this arm | NA (NA) — no participants with data on this day in this arm | 11.0 (24.04) | 3.3 (4.62)
  QRS at Day 113 (n=0,0,2,3) | NA (NA) — no participants with data on this day in this arm | NA (NA) — no participants with data on this day in this arm | 4.0 (2.83) | 6.0 (6.93)
  QT at Day 113 (n=0,0,2,3) | NA (NA) — no participants with data on this day in this arm | NA (NA) — no participants with data on this day in this arm | 4.0 (50.91) | 6.0 (28.00)

17. Secondary Outcome: Mean Diastolic Blood Pressure at Baseline and Post-Infusion Day 1 (Cycle 1) in 0.3 mg Cohort - Safety Population
Description: Diastolic blood pressures (DBPs) measured in millimeters of mercury (mmHg) were obtained while the participant was seated. Post infusion DBPs are presented in the 0.3 mg cohort at: 21, 36, 51, 66, 82, 97, 112, 127, 157 minutes post infusion, and at 1, 2, 3, 4, 6, 8 hours post infusion. Baseline was defined as the last measurement before the first dose of study drug, which was calculated from pre-dose or from screening if pre-dose was not available. Mean DBP on Day 1 for first dose (cycle 1) are presented below.
Time Frame: Baseline, Day 1
Population: All participants who received at least 1 dose or any partial dose of nivolumab and had available blood pressure at baseline and post-infusion were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 0.3 mg/kg Nivolumab
Number analyzed (Participants) | 6
mmHg
  Baseline (n=6) | 80.3 (18.16)
  Infusion (0 minutes) (n=5) | 82.4 (10.01)
  21 minutes post infusion (n=6) | 87.0 (10.28)
  36 minutes post infusion (n=6) | 81.0 (10.88)
  51 minutes post infusion (n=6) | 79.8 (9.20)
  66 minutes post infusion (n=6) | 80.3 (8.71)
  82 minutes post infusion (n=6) | 81.7 (8.69)
  97 minutes post infusion (n=6) | 80.3 (10.56)
  112 minutes post infusion (n=6) | 78.7 (8.14)
  127 minutes post infusion (n=6) | 81.0 (11.14)
  157 minutes post infusion (n=2) | 72.5 (6.36)
  1 hour post infusion (n=6) | 80.5 (8.96)
  2 hour post infusion (n=6) | 82.2 (11.02)
  3 hour post infusion (n=6) | 74.5 (6.35)
  4 hour post infusion (n=6) | 73.8 (6.08)
  6 hour post infusion (n=6) | 78.2 (10.44)
  8 hour post infusion (n=6) | 76.2 (5.67)

18. Secondary Outcome: Mean Systolic Blood Pressure at Baseline and Post-Infusion Day 1 (Cycle 1) in 0.3 mg Cohort - Safety Population
Description: Systolic blood pressures (SBPs) measured in millimeters of mercury (mmHg) were obtained while the participant was seated. Baseline, Infusion (0 minutes) and Post infusion SBPs are presented in the 0.3 mg cohort at: 21, 36, 51, 66, 82, 97, 112, 127, 157 minutes post infusion, and at 1, 2, 3, 4, 6, 8 hours post infusion. Baseline was defined as the last measurement before the first dose of study drug, which was calculated from pre-dose or from screening if pre-dose was not available. Mean SBP on Day 1 for first dose (cycle 1) are presented below.
Time Frame: Baseline, Day 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 0.3 mg/kg Nivolumab
Number analyzed (Participants) | 6
mmHg
  Baseline (n=6) | 141.8 (15.03)
  Infusion (0 minutes) (n=5) | 144.2 (17.05)
  21 minutes post infusion (n=6) | 154.3 (22.90)
  36 minutes post infusion (n=6) | 140.3 (14.71)
  51 minutes post infusion (n=6) | 147.5 (10.05)
  66 minutes post infusion (n=6) | 141.0 (15.44)
  82 minutes post infusion (n=6) | 145.7 (17.60)
  97 minutes post infusion (n=6) | 141.8 (16.29)
  112 minutes post infusion (n=6) | 139.8 (11.55)
  127 minutes post infusion (n=6) | 140.3 (20.47)
  157 minutes post infusion (n=2) | 137.5 (7.78)
  1 hour post infusion (n=6) | 139.3 (8.04)
  2 hour post infusion (n=6) | 145.8 (20.85)
  3 hour post infusion (n=6) | 140.3 (7.92)
  4 hour post infusion (n=6) | 139.8 (9.89)
  6 hour post infusion (n=6) | 142.8 (19.06)
  8 hour post infusion (n=6) | 145.5 (12.77)

19. Secondary Outcome: Mean Diastolic Blood Pressure at Baseline and Post-Infusion Day 1 (Cycle 1) in 1mg, 3mg, and 10 mg Cohorts - Safety Population
Description: Diastolic blood pressures (DBPs) measured in millimeters of mercury (mmHg) were obtained while the participant was seated. Baseline, Infusion (0 minutes) and Post infusion DBPs are presented in the 1 mg, 3 mg and 10 mg cohorts at: 15, 30, 45, 60, 75, and 90 minutes post infusion and at 1, 2, 3, 4, 6, 8 hours post infusion. Baseline was defined as the last measurement before the first dose of study drug, which was calculated from pre-dose or from screening if pre-dose was not available. Mean DBP on Day 1 for first dose (cycle 1) are presented below.
Time Frame: Baseline, Day 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 6 | 6 | 21
mmHg
  Baseline (n=6, 6, 21) | 80.3 (11.62) | 72.2 (10.72) | 74.4 (12.19)
  Infusion (0 minutes) (n=6, 5, 19) | 79.2 (11.72) | 73.6 (10.01) | 74.2 (11.31)
  15 minutes post infusion (n=6,6,21) | 74.5 (11.41) | 69.5 (10.41) | 72.3 (11.87)
  30 minutes post infusion (n=6,6,21) | 78.8 (11.0) | 70.7 (10.29) | 71.1 (10.40)
  45 minutes post infusion (n=6,6,21) | 75.7 (10.67) | 69.8 (12.09) | 72.7 (12.69)
  60 minutes post infusion (n=6,6,21) | 78.7 (8.78) | 69.5 (9.97) | 74.1 (10.53)
  75 minutes post infusion (n=5,3,12) | 79.0 (11.20) | 71.7 (0.58) | 73.7 (11.93)
  90 minutes post infusion (n=4,4,14) | 79.8 (8.73) | 70.3 (8.18) | 74.4 (11.09)
  1 hour post infusion (n= 6,5,21) | 78.5 (7.58) | 74.4 (17.18) | 71.9 (10.24)
  2 hour post infusion (n= 6,6,21) | 83.0 (10.35) | 70.7 (19.04) | 72.0 (10.62)
  3 hour post infusion (n= 6,5,19) | 79.5 (13.20) | 67.8 (24.59) | 72.9 (11.98)
  4 hour post infusion (n= 6,6,21) | 75.2 (17.68) | 69.2 (13.64) | 73.5 (9.86)
  6 hour post infusion (n= 6,6,21) | 74.7 (7.81) | 77.7 (13.35) | 73.1 (10.32)
  8 hour post infusion (n= 5,5,21) | 83.8 (8.04) | 76.4 (15.29) | 74.7 (8.33)

20. Secondary Outcome: Mean Systolic Blood Pressure at Baseline and Post-Infusion Day 1 (Cycle 1) in in 1mg, 3mg, and 10 mg Cohorts - Safety Population
Description: Systolic blood pressures (SBPs) measured in millimeters of mercury (mmHg) were obtained while the participant was seated. Baseline, Infusion (0 minutes) and Post infusion SBPs are presented in the 1 mg, 3 mg and 10 mg cohorts at: 15, 30, 45, 60, 75, and 90 minutes post infusion and at 1, 2, 3, 4, 6, 8 hours post infusion. Baseline was defined as the last measurement before the first dose of study drug, which was calculated from pre-dose or from screening if pre-dose was not available. Mean SBPs on Day 1 for first dose (cycle 1) are presented below.
Time Frame: Baseline, Day 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 6 | 6 | 21
mmHg
  Baseline (n=6, 6, 21) | 133.2 (2.86) | 121.3 (13.11) | 128.8 (19.29)
  Infusion (0 minutes) (n=6, 5, 19) | 138.8 (10.65) | 116.4 (8.56) | 129.5 (17.38)
  15 minutes post infusion (n=6,6,21) | 136.7 (12.03) | 117.3 (8.64) | 125.5 (16.54)
  30 minutes post infusion (n=6,6,21) | 139.2 (6.71) | 119.8 (10.82) | 124.0 (14.00)
  45 minutes post infusion (n=6,6,21) | 141.2 (12.19) | 111.5 (5.79) | 123.5 (14.38)
  60 minutes post infusion (n=6,6,21) | 142.3 (3.78) | 115.0 (5.69) | 124.8 (14.39)
  75 minutes post infusion (n=5,3,12) | 134.0 (8.69) | 119.3 (10.21) | 126.2 (18.01)
  90 minutes post infusion (n=4,4,14) | 134.0 (7.62) | 119.0 (8.76) | 126.1 (14.24)
  1 hour post infusion (n= 6,5,21) | 141.2 (5.74) | 120.6 (15.69) | 121.2 (16.72)
  2 hour post infusion (n= 6,6,21) | 131.3 (9.91) | 119.7 (11.04) | 123.4 (14.76)
  3 hour post infusion (n= 6,5,19) | 133.5 (9.79) | 122.2 (12.24) | 125.4 (15.29)
  4 hour post infusion (n= 6,6,21) | 133.0 (9.94) | 128.5 (19.61) | 125.9 (13.20)
  6 hour post infusion (n= 6,6,21) | 137.0 (11.63) | 130.0 (14.21) | 124.6 (15.77)
  8 hour post infusion (n= 5,5,21) | 144.8 (13.81) | 130.6 (19.36) | 130.6 (12.21)

ADVERSE EVENTS:
Time Frame: Day 1 through long-term follow-up until either progressive disease or 2 years elapsed.
Description: Study was initiated in 2006 and completed in 2009
Groups:
- 0.3 mg/kg Nivolumab: 0.3 mg of nivolumab per kg of body weight was administered in a single IV infusion on Day 1 with 10% of the dose infused over 6 minutes and after a 1 hour observation period, the balance was administered over 60 minutes. Eligible participants could be re-treated and receive 2 more doses (1 dose every 4 weeks) at same dose as the single dose if: disease was stable, no drug intolerance was observed, no complete response (CR) or partial response (PR) was observed, or they had a positive immunogenicity sample within 4 weeks prior to re-treatment. Those who responded to therapy with a CR or PR were eligible for long-term follow-up until either progressive disease (PD) or 2 years elapsed.
Arm/Group | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Serious Adverse Events (participants affected / at risk) | 3/6 | 5/6 | 4/6 | 11/21
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.3 mg/kg Nivolumab (N=6) | 1 mg/kg Nivolumab (N=6) | 3 mg/kg Nivolumab (N=6) | 10 mg/kg Nivolumab (N=21)
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 1 | 4
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bladder obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.3 mg/kg Nivolumab (N=6) | 1 mg/kg Nivolumab (N=6) | 3 mg/kg Nivolumab (N=6) | 10 mg/kg Nivolumab (N=21)
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 2 | 3 | 1 | 3
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 9
Blood chloride decreased (Investigations) | 0 | 1 | 1 | 1
Blood thyroid stimulating hormone increased (Investigations) | 1 | 1 | 1 | 4
Carbon dioxide decreased (Investigations) | 0 | 4 | 4 | 6
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 2
Crystal urine present (Investigations) | 0 | 1 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Electrocardiogram ST-T change (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Glucose urine (Investigations) | 0 | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 4 | 3 | 8
Hypotension (Vascular disorders) | 0 | 0 | 0 | 3
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 1 | 4
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 9
Weight decreased (Investigations) | 5 | 2 | 3 | 9
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 0 | 4
Blood uric acid decreased (Investigations) | 0 | 0 | 0 | 2
CD4 lymphocytes decreased (Investigations) | 1 | 2 | 1 | 14
Crystal urine (Investigations) | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 1 | 0 | 0 | 2
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 2 | 7
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Eosinophil count increased (Investigations) | 0 | 1 | 0 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 5
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 4
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
T-lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 4
Tachycardia (Cardiac disorders) | 2 | 1 | 0 | 3
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 4
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
B-lymphocyte count increased (Investigations) | 0 | 0 | 1 | 0
Bacteria urine (Investigations) | 0 | 1 | 0 | 1
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 5
Blood creatinine increased (Investigations) | 0 | 2 | 2 | 1
Blood phosphorus increased (Investigations) | 0 | 1 | 3 | 3
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 1
Blood urine present (Investigations) | 1 | 0 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Eosinophil count decreased (Investigations) | 1 | 2 | 0 | 4
Eye pain (Eye disorders) | 0 | 1 | 1 | 0
Haematocrit decreased (Investigations) | 1 | 1 | 0 | 2
Haemoglobin decreased (Investigations) | 2 | 4 | 1 | 4
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypergammaglobulinaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 3 | 2 | 5
Influenza like illness (General disorders) | 0 | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 4
Mean cell volume decreased (Investigations) | 1 | 0 | 0 | 3
Monocyte count increased (Investigations) | 0 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 2
Pruritus ani (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0
Rheumatoid factor (Investigations) | 0 | 0 | 1 | 0
Rheumatoid factor positive (Investigations) | 0 | 0 | 0 | 3
White blood cell count increased (Investigations) | 2 | 1 | 1 | 3
White blood cells urine (Investigations) | 0 | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 3 | 12
Blood bicarbonate decreased (Investigations) | 1 | 4 | 3 | 5
Blood bilirubin increased (Investigations) | 0 | 2 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 2 | 1 | 4
Blood magnesium decreased (Investigations) | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 4 | 4 | 8
Catheter site erythema (General disorders) | 0 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 2 | 1 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 4
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 2
Protein total decreased (Investigations) | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 7
Scrotal swelling (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Thyroxine decreased (Investigations) | 0 | 0 | 2 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 2
Urine colour abnormal (Investigations) | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 2 | 0 | 1
B-lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 4
Blood sodium decreased (Investigations) | 0 | 1 | 0 | 5
Blood urea decreased (Investigations) | 1 | 1 | 0 | 1
CD8 lymphocytes decreased (Investigations) | 1 | 1 | 0 | 1
Carbon dioxide increased (Investigations) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2 | 6
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 7
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Infusion site oedema (General disorders) | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Monocyte count decreased (Investigations) | 1 | 0 | 0 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Neutrophil count increased (Investigations) | 1 | 2 | 1 | 5
Oedema (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 2 | 3 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Pyrexia (General disorders) | 1 | 2 | 2 | 4
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Urinary sediment present (Investigations) | 1 | 3 | 1 | 7
Apraxia (Nervous system disorders) | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 2 | 0 | 6
Asthenia (General disorders) | 1 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 2 | 3 | 13
Breath sounds abnormal (Investigations) | 0 | 1 | 0 | 0
CD4 lymphocytes increased (Investigations) | 0 | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 5
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 5 | 4 | 12
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 0 | 0
Hypochromasia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 2
Mean cell haemoglobin concentration decreased (Investigations) | 0 | 2 | 0 | 4
Microcytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 4 | 11
Proteinuria (Renal and urinary disorders) | 2 | 3 | 2 | 8
Red blood cell count decreased (Investigations) | 1 | 1 | 0 | 1
Red blood cells urine (Investigations) | 0 | 0 | 0 | 3
Rheumatoid factor increased (Investigations) | 0 | 1 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 3
Specific gravity urine increased (Investigations) | 1 | 1 | 1 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 3
White blood cells urine positive (Investigations) | 0 | 1 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 3 | 1 | 4
Blood calcium decreased (Investigations) | 0 | 2 | 0 | 3
Blood chloride increased (Investigations) | 0 | 0 | 1 | 3
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 2 | 0
Blood glucose increased (Investigations) | 0 | 1 | 1 | 7
Blood urea increased (Investigations) | 1 | 3 | 0 | 3
Blood uric acid increased (Investigations) | 1 | 2 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 3
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 5
Facial wasting (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Gait disturbance (General disorders) | 0 | 0 | 1 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2 | 2 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 4 | 1 | 3 | 9
Mean cell haemoglobin decreased (Investigations) | 1 | 1 | 0 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Platelet count increased (Investigations) | 3 | 1 | 1 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Antinuclear antibody positive (Investigations) | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2
Blood phosphorus decreased (Investigations) | 1 | 1 | 0 | 2
Blood potassium increased (Investigations) | 0 | 0 | 0 | 3
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 2 | 1 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 3 | 10
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Interleukin level increased (Investigations) | 0 | 2 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 3 | 1 | 6
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Thyroxine free increased (Investigations) | 0 | 0 | 1 | 1
White blood cell count decreased (Investigations) | 2 | 1 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.